CLINICAL TRIAL: NCT03110497
Title: A Feasibility and Safety Study of Single Application Multi-fractionated High Dose Rate (HDR) Brachytherapy in Locally Advanced Cervical Cancer
Brief Title: Single Application Brachytherapy in Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Umesh Mahantshetty, Professor, Tata Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMH-1759; REF/2017/03/013733 (Registry Identifier: Clinical Trial Registry - India)
Record Dates: First submitted 2017-03-24; First posted 2017-04-12 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-01

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; Image guided Brachytherapy; single application
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase I/ Phase II single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single application brachytherapy (Experimental): After external beam radiotherapy with or without chemotherapy as per standard, each study patient will undergo single application brachytherapy to deliver 3 High Dose Rate (HDR) fractions [1st, 2nd and 3rd fractions of doses 9 Gy, 7 Gy and 7 Gy respectively] keeping 6-12 hours of interval. All patients will undergo an inter-fraction Computed Tomography (CT) scan before delivery of second fraction. Plan will be re-optimized to reduce the dose to Organs at Risk (OAR's), only if the dose exceeds the dose constraints. Dose constraints being exceedingly hard in 1st fraction or before 2nd fraction even after re-planning will deem patient non-feasible but optimization will be done to give preference to OAR's while accepting some compromise in target doses.
  Interventions: Radiation: Single application multi-fraction brachytherapy

INTERVENTIONS:
Radiation: Single application multi-fraction brachytherapy — Single application brachytherapy procedure to deliver high dose rate fractions of 9Gy, 7Gy and 7Gy with 6-12 hours apart under strict image guidance

SUMMARY:
The purpose of the study is to evaluate safety and feasibility of single brachytherapy application with dose delivery in multiple fractions. Study will be conducted in Phase I/II clinical trial setting with strict Image guidance protocol.This study is expected reduce treatment duration and to increase ease and acceptability of brachytherapy in patients along with significant saving of resources

DETAILED DESCRIPTION:
Brachytherapy for cervical cancers has evolved a long way from the era of Manchester based point A prescription to volume-based prescription in the current era of 3 Dimensional (3D) imaging. Advancement in imaging technology and widespread availability of this technology has allowed most centers worldwide to incorporate Image guided brachytherapy as a routine part of their clinical practice.

The primary advantage of 3D image guided brachytherapy is that it allows the dose given by brachytherapy to conform to the anatomy of each individual patient while reducing the doses to organs at risk (OAR) (1). This technique has shown to improve local control rates and also reduce the rates of moderate to severe morbidity in multiple single institutional series (2-6). However, treatment related urinary and gastrointestinal late morbidity is still a significant problem with the 3 year actuarial incidence of intermediate to major morbidity (Grade≥2) being 30% and 29% for urinary and gastrointestinal side effects, respectively and Major morbidity (Grade≥3) is seen in 7% and 8%, respectively [An intErnational study on MRI guided BRachytherapy in locally Advanced CErvical cancers (EMBRACE) study 2014, work in progress(7)].

Most important factor determining late toxicities in radiotherapy is dose per fraction and total dose (total BEDGy3) rather than rate of dose accumulation or number of applications, which is evident from many trials of HDR brachytherapy.

The dose per fraction in the protocol of 9Gy, 7Gy and 7Gy HDR is effective in terms of local control rates and toxicities which has been published(8,9).

Our study is designed to evaluate the feasibility to deliver complete course of HDR brachytherapy in a single application while achieving dose constraints to OARs and keeping in account inter-fraction variation of doses to OAR's.

In the protocol proposed here, The Investigators intend to deliver fractionated treatments in a strict image based and quality controlled environment to minimize the doses to OAR's. Also if the constraints are not achieved, patients would be offered Standard brachytherapy regimen. This would ensure that the anticipated late toxicities would be minimized.

This study is expected to decrease overall treatment time and increase the ease and acceptability of brachytherapy in patients and with significant saving of resources while maintaining disease control rates and toxicity rates similar to standard protocols.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed invasive cervical cancer (squamous carcinoma, adenosquamous carcinoma, adenocarcinoma)
* International Federation of Gynecology and Obstetrics (FIGO) stage 2b-4a after thorough clinical examination and work-up investigation
* Suitable for radical radiation therapy with/without chemotherapy, and also for brachytherapy boost
* Accepts the Informed consent process and signs the form on his/her will.

Exclusion Criteria:

* Patients with vesico-vaginal fistula or recto-vaginal fistula at diagnosis
* Patients at high risk of anaesthesia and patients with phobia /contra-indications to undergo MRI
* Patients not suitable for brachytherapy
* Metastatic disease beyond iliac on standard imaging
* Vault cancers/recurrence
* Previous history of pelvic radiation
* Non-compliance to treatment
* Medical or psychological illness precluding treatment protocol

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Study conducted for females with cervical cancer
Enrollment: 40 (Estimated)
Dates: Start 2017-09-17 (Actual); Primary Completion 2019-04-17 (Estimated); Study Completion 2020-04-17 (Estimated)

PRIMARY OUTCOMES:
Number of participants achieving specified dosimetric constraints | 1 year
  Number of participants achieving protocol specified dosimetric constraints will be measured, these dosimetric constraints are considered as a measure of safety. If not more than 20% of participants fail to achieve dosimetric constraints, trial will be considered feasible.

SECONDARY OUTCOMES:
Number of participants with adverse events as assessed by CTCAE v 4.0 | 2 years
  To assess toxicity outcomes in terms of treatment related late Gastrointestinal (GI) / Genitourinary (GU) / Vaginal toxicities (grade 3 or more)
Local control rate | 2 years
  Status of local disease at 2 years after treatment
Percentage Inter-fraction dose variation | 1 year
  To evaluate inter fraction dose variation for organs at risk

CONTACTS AND LOCATIONS:
Overall Officials: Umesh Mahantshetty, MD, DNB, Principal Investigator — Professor, Department of Radiation oncology, Tata memorial Centre, Mumbai
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tanderup K, Nielsen SK, Nyvang GB, Pedersen EM, Rohl L, Aagaard T, Fokdal L, Lindegaard JC. From point A to the sculpted pear: MR image guidance significantly improves tumour dose and sparing of organs at risk in brachytherapy of cervical cancer. Radiother Oncol. 2010 Feb;94(2):173-80. doi: 10.1016/j.radonc.2010.01.001. PMID 20138380
- [Background] Lindegaard JC, Fokdal LU, Nielsen SK, Juul-Christensen J, Tanderup K. MRI-guided adaptive radiotherapy in locally advanced cervical cancer from a Nordic perspective. Acta Oncol. 2013 Oct;52(7):1510-9. doi: 10.3109/0284186X.2013.818253. Epub 2013 Aug 21. PMID 23962242
- [Background] Potter R, Dimopoulos J, Georg P, Lang S, Waldhausl C, Wachter-Gerstner N, Weitmann H, Reinthaller A, Knocke TH, Wachter S, Kirisits C. Clinical impact of MRI assisted dose volume adaptation and dose escalation in brachytherapy of locally advanced cervix cancer. Radiother Oncol. 2007 May;83(2):148-55. doi: 10.1016/j.radonc.2007.04.012. PMID 17531904
- [Background] Potter R, Georg P, Dimopoulos JC, Grimm M, Berger D, Nesvacil N, Georg D, Schmid MP, Reinthaller A, Sturdza A, Kirisits C. Clinical outcome of protocol based image (MRI) guided adaptive brachytherapy combined with 3D conformal radiotherapy with or without chemotherapy in patients with locally advanced cervical cancer. Radiother Oncol. 2011 Jul;100(1):116-23. doi: 10.1016/j.radonc.2011.07.012. Epub 2011 Aug 5. PMID 21821305
- [Background] Sturdza A, Potter R, Fokdal LU, Haie-Meder C, Tan LT, Mazeron R, Petric P, Segedin B, Jurgenliemk-Schulz IM, Nomden C, Gillham C, McArdle O, Van Limbergen E, Janssen H, Hoskin P, Lowe G, Tharavichitkul E, Villafranca E, Mahantshetty U, Georg P, Kirchheiner K, Kirisits C, Tanderup K, Lindegaard JC. Image guided brachytherapy in locally advanced cervical cancer: Improved pelvic control and survival in RetroEMBRACE, a multicenter cohort study. Radiother Oncol. 2016 Sep;120(3):428-433. doi: 10.1016/j.radonc.2016.03.011. Epub 2016 Apr 29. PMID 27134181
- [Background] Fokdal L, Sturdza A, Mazeron R, Haie-Meder C, Tan LT, Gillham C, Segedin B, Jurgenliemk-Schultz I, Kirisits C, Hoskin P, Potter R, Lindegaard JC, Tanderup K. Image guided adaptive brachytherapy with combined intracavitary and interstitial technique improves the therapeutic ratio in locally advanced cervical cancer: Analysis from the retroEMBRACE study. Radiother Oncol. 2016 Sep;120(3):434-440. doi: 10.1016/j.radonc.2016.03.020. Epub 2016 Apr 21. PMID 27113795
- [Background] Patel FD, Sharma SC, Negi PS, Ghoshal S, Gupta BD. Low dose rate vs. high dose rate brachytherapy in the treatment of carcinoma of the uterine cervix: a clinical trial. Int J Radiat Oncol Biol Phys. 1994 Jan 15;28(2):335-41. doi: 10.1016/0360-3016(94)90055-8. PMID 8276647
- [Background] Shrivastava S DK, Mahantshetty U, Engineer R, Patil N, Deshpande D, Tongaonkar H Comparing Low-Dose-Rate andHigh-Dose-Rate Intracavitary Brachytherapy in Carcinoma Cervix: Results From a Randomized Controlled Study. . Int J Radiat Oncol Biol Phys 2006, 1; 66.
- See also: EMBRACE Study — http://www.embracestudy.dk